CLINICAL TRIAL: NCT01638702
Title: Assessment of Impact of Choice of Arm for Access on Rate of Complications in Peripherally Inserted Central Venous Catheters
Brief Title: Study of Complication Rates Associated With PICC for Left vs Right
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Lindsay (Other)
Responsible Party: Sponsor-Investigator, Richard Lindsay, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-086-BMB
Record Dates: First submitted 2012-06-18; First posted 2012-07-12 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Bacterial Infections
Keywords: Catheterisation, Central Venous; Catheters, Indwelling
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right sided PICC placement (Active Comparator): Insertion of PICC on the right arm
  Interventions: Other: Follow up of complications
- Left sided arm placement (Placebo Comparator): Insertion of PICC on the left arm
  Interventions: Other: Follow up of complications

INTERVENTIONS:
Other: Follow up of complications — Follow up for complications leading or not to removal (occlusion, accidental removal, infection, catheter related thrombosis, leaking, pain...)

SUMMARY:
Peripherally inserted central catheter (PICC) are catheters that are placed mainly in the arms, but which pass in the veins to beside the heart. They are associated with occasional complications due to infection or blockage of the vein that they are in. The investigators want to investigate whether PICCs in the right arm have lower complications than those in the left. This difference in complication rates has been noticed in most other forms of central venous access.

ELIGIBILITY:
Inclusion Criteria:

* Referral for in-patient PICC placement at centre carrying out study.

Exclusion Criteria:

* Out of hospital referrals for PICC placement; previous PICC placement; previous long term central catheter/pacemaker; unable to give valid consent; presence of pre-existing medical preventing randomisation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Line infection rate | From insertion to line removal, an estimated time of 4 weeks
  All patients will be followed from the point of time of randomisation and PICC insertion until the line develops a complication or is removed. The average length of duration of line access in our institution is 4 weeks.

SECONDARY OUTCOMES:
Effect of number of lumens | From insertion to time of removal, an estimated average time of four weeks.
  Assessing the effect number of lumens in the catheter has on complication rate.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lindsay, MB Bch BaO, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; France Paquet, BS(N) MS(N), Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided